CLINICAL TRIAL: NCT06290778
Title: Peer Delivered, Emotion Regulation-Focused Mental Health Prevention Training for Fire Fighter Trainees
Acronym: PEER UP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: University of Pittsburgh (Other); Boston University (Other); Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Baylor IRB #023-445
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: PTSD; Alcohol Use Disorder; Depression; Anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Unified Protocol (Experimental): This workshop includes education regarding basic human emotions, why we have emotions, how they help us, how they can get in the way, and how they are related to psychological health problems, including among firefighters. Skills that are helpful in managing strong or unwanted emotions will be taught and practiced during the workshop. A workshop manual will be provided. Brief videos summarizing the material will be emailed over the course of the month following the workshop.
  Interventions: Behavioral: Brief Unified Protocol
- Psychoeducation (Active Comparator): This workshop provides education regarding signs and symptoms of psychological health challenges that are most commonly experienced by firefighters. These include posttraumatic stress, depression, anxiety, and alcohol and substance misuse. This workshop is a standard part of fire academy training. A workshop manual will be provided. Brief videos summarizing the material will be emailed over the course of the month following the workshop.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Brief Unified Protocol — The Brief Transdiagnostic Treatment of Emotional Disorders Unified Protocol.
  Arms: Brief Unified Protocol
Behavioral: Psychoeducation — Psychoeducation regarding mental health challenges in fire service.
  Arms: Psychoeducation

SUMMARY:
The goal of this clinical trial is to determine if a peer-delivered emotion regulation training (Brief-Unified Protocol) workshop is effective for preventing posttraumatic stress and other psychological health symptoms in firefighter trainees. The main questions it aims to answer are:

* Do firefighter recruits who receive peer-delivered Brief-Unified Protocol report lower PTSD symptom severity over time compared to those who receive psychoeducation?
* Do firefighter recruits who receive peer-delivered Brief-Unified Protocol report lower AUD, depression, anxiety, and functional impairment symptom severity over time compared to those who receive psychoeducation?
* Do changes in neuroticism or emotion regulation mediate the effect of receiving the Brief-Unified Protocol on the treatment outcomes?

Participants will:

* Participate in a Brief-Unified Protocol workshop or psychoeducation workshop during fire academy training.
* Complete a questionnaire prior to the workshop.
* Complete a questionnaire immediately following the workshop and follow up questionnaires at 6, 12, 18, and 24 months after completing the fire academy.

Researchers will compare firefighters who receive a peer-delivered Brief-Unified Protocol workshop to firefighters who receive peer-delivered psychoeducation to see if the Brief-Unified Protocol is effective for preventing posttraumatic stress and other psychological health symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* English speaking
* Able to sign an informed consent form
* Able to complete the self-report assessment
* Willing to be contacted to complete post and follow-up assessments

Exclusion Criteria:

* Pregnant
* Have plans to relocate within two months of protocol initiation
* Report psychotic symptoms or suicidal behavior within the past 2 weeks
* Are currently dependent on substances other than tobacco or caffeine

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptoms | 6, 12, 18, and 24 months
  PTSD Checklist-5 (PCL-5). Score Range: 0-80. Higher scores indicate greater severity.

SECONDARY OUTCOMES:
Alcohol Use Disorder symptoms | 6, 12, 18, and 24 months
  Alcohol Use Disorders Identification Test (AUDIT). Score Range: 0-40. Higher scores indicate a higher likelihood of alcohol dependence.
Depression symptoms | 6, 12, 18, and 24 months
  Patient Health Questionnaire (PHQ-9). Score Range: 0-27. Higher scores indicate greater severity.
Anxiety symptoms | 6, 12, 18, and 24 months
  Generalized Anxiety Disorder (GAD-7). Score Range: 0-21. Higher scores indicate greater severity.
Functional Impairment | 6, 12, 18, and 24 months
  Work and Social Adjustment Scale (WSAS). Score Range: 0-40. Higher scores indicate greater functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- MacArthur Clinic, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer EC, Farchione T, Kimbrel NA, Kwok OM, Pennington ML, Rostockyj J, Gulliver SB. Peer delivered, emotion regulation-focused mental health prevention training for fire fighter trainees: Design and methodology of a randomized controlled trial. Contemp Clin Trials Commun. 2025 Aug 18;47:101537. doi: 10.1016/j.conctc.2025.101537. eCollection 2025 Oct. PMID 40893729